CLINICAL TRIAL: NCT06249269
Title: Reversal of Atrial Substrate to Prevent Atrial Fibrillation Cohort Study
Acronym: RASTA-Cohort
Status: Recruiting | Type: Observational
Sponsor: Ratika Parkash (Other)
Collaborators: Nova Scotia Health Research Fund (Unknown)
Responsible Party: Sponsor-Investigator, Ratika Parkash, Physician, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: RP-08
Record Dates: First submitted 2024-01-03; First posted 2024-02-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation, Paroxysmal or Persistent
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RASTA AF Cohort: Patients who meet the inclusion criteria for RASTA-AF, and do not meet any of the exclusion criteria but decline or are not approached for participation in the RCT will be asked to participate.

SUMMARY:
Atrial fibrillation (AF) is a major health problem, with a prevalence of 0.4-1% of the population. It results in high healthcare costs and significant morbidity, especially for patients with severe symptoms. The RASTA-AF randomized control trial (RCT) is designed to answer the following question: does vigorous treatment of AF with aggressive risk factor management plus catheter ablation reduce AF-related outcomes as compared to catheter ablation plus usual care in patients with symptomatic AF and risk factors that promote AF.

This study is a multicenter, prospective cohort study that will enrol patients who decline participation in the RASTA-AF RCT but agree to be followed in a registry. The objective of RASTA-Cohort is to determine whether patients who decline participation in the RASTA-AF RCT have different clinical characteristics and quality of life than patients who accept participation in the study, and whether they suffer from worse AF-related outcomes than patients in the RCT.

DETAILED DESCRIPTION:
Randomized clinical trials remain the gold standard for determining the efficacy of an intervention, however, it is well known that patients will decline participation in clinical trials for various reasons. It is critical to understand outcomes of patients who are eligible for a clinical trial, but decline participation, as it may affect the magnitude of an intervention, and ultimately its clinical meaningfulness. The RASTA cohort study will address this issue in patients with AF. Atrial fibrillation has become a significant burden globally, and is more often present in older individuals. This is particularly important in Nova Scotia where our healthcare system is especially burdened as the population ages, 20% of the current population is >65 years. Improved understanding of the AF patient population in Nova Scotia, and beyond, will permit further understanding of how best to treat this increasingly common chronic illness.

The RASTA-Cohort study is designed to answer the following questions:

1. Do patients who decline participation in the RASTA AF RCT have different clinical characteristics and quality of life than patients who accept participation in the study.
2. Do patients who do not participate in the RASTA AF RCT suffer from worse AF-related outcomes than patients in the study, as compared to the control arm and intervention arm.

This is a multicenter, prospective cohort study that will enrol patients who are eligible for, but do not participate in the RASTA-AF study, but agree to be followed in this registry. Once the patient has consented to participate in RASTA Cohort, they will be scheduled for their AF ablation at the next available timeframe (2-4 months from entry into the study). All patients will continue to receive care as per current guidelines; this will be managed at the discretion of their treating physician.

Clinical characteristics collected at baseline include quality of life (CCS-SAF, AFEQT, EQ-5D), physical activity measures: IPAQ and stress test results (where available), blood pressure, weight, hemoglobin A1C, alcohol use and smoking cessation. The measures of risk factors will be performed in a similar fashion as the main study to ensure that these can be compared.

The conservative estimated event rate for the cohort is 20% greater than that of the control population of the RASTA AF study. Given the control population having an event rate of 30%, and the cohort group being 43.5%, a sample size of 313 patients is required in the control population of RASTA and 185 patients in the cohort group with a minimum 2 year follow up. Using a 7% loss to follow up rate, the sample size required in the cohort group is 198 patients. This sample size will provide 90% power with a type I error of 0.05 to detect a difference in survival between the cohort and the control group in the study. There is >99% power to detect a difference between the intervention group and the cohort group based on the sample of 198 patients.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic AF (CCS-SAF ≥2),
* paroxysmal or persistent atrial fibrillation despite rate control, desiring catheter ablation and either: i) BMI ≥ 30 or, ii) at least two of the following: BMI>27, BP>140/90 mmHg or history of hypertension, Diabetes, Heart failure (prior heart failure admission or LVEF<40%), Age ≥ 65 years, Prior stroke/TIA, Current smoker, Excessive alcohol use {For women: 10 or more drinks/week, more than 2 drinks a day (most days). For men: 15 or more drinks/week, more than 3 drinks a day (most days)}, and iii) declined or were not approached for participation in the main study. Eligible patients must have received catheter ablation for AF during the same timeline of the RASTA-AF Mian Study (November 1st, 2019 to December 31st, 2025).

Exclusion Criteria:

* permanent AF (AF lasting > 3 years),
* prior catheter ablation for AF
* New York Heart Association Class IV heart failure
* participation in a cardiac rehabilitation program within the last year,
* currently performing exercise training >150 minutes/week of moderate to vigorous physical activity,
* unable to exercise,
* unable to give informed consent,
* other noncardiovascular medical condition making 1 year survival unlikely
* less than 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with persistent or paroxysmal AF requiring catheter ablation and meet the inclusion/exclusion criteria for RASTA-AF, but decline or are not approached for participation in the Randomized Clinical Trial will be asked to participate in RASTA Cohort.
Sampling Method: Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with atrial fibrillation (AF) related hospitalizations | Up to 60 months
  Defined as any hospitalization (greater than 24 hours) from 2 months post ablation to end of follow up due to: atrial fibrillation/atrial flutter, stroke/transient ischemic attack/systemic embolism, heart failure, syncope or bradycardia requiring pacing.
Number of patients with atrial fibrillation (AF) related ED visits | Up to 60 months
  Defined as any presentation to the emergency department (less than 24 hours) due to: atrial fibrillation/atrial flutter, stroke/transient ischemic attack/systemic embolism, heart failure, syncope or bradycardia requiring pacing.
Number of patients with clinically significant atrial fibrillation post ablation | Up to 60 months
  Clinically significant AF events lasting greater or equal to 24 hours within 26 hours (either an irregular R-R interval or atrial cycle length less than 280 ms, as obtained from an insertable cardiac monitor) from 2 months post ablation to end of follow-up.

SECONDARY OUTCOMES:
Number of patients with a composite of AF-related hospitalizations and ED visits or clinically significant AF | Up to 60 months
  Defined as any hospitalization or presentation to the emergency department due to: atrial fibrillation/atrial flutter, stroke/transient ischemic attack/systemic embolism, heart failure, syncope or bradycardia requiring pacing and/or clinically significant atrial fibrillation (greater than or equal to 24 hours with symptoms) from randomization to end of follow up.
Number of patients with stroke or systemic embolism | Up to 60 months
  Hospitalization or treatment for a stroke or systemic embolism
Quality of Life - CCS SAF scale | Up to 60 months
  Symptom burden as measured by the Canadian Cardiovascular Society (CCS) Severity of Atrial Fibrillation (SAF) Scale. CCS-SAF scores range from 0 to 4, with higher values representing more severe impact of AF-related symptoms on quality of life and activities of daily living.
Quality of Life - AFEQT | Up to 60 months
  Quality of life scale as measured by the Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) scale. The scale consists of 21 questions with 7-point Likert scale responses. Questions 1-18 are grouped into three subscales (symptoms, daily activities and treatment concern). Questions 19-21 capture satisfaction with treatment and are not included in the HRQoL score of the questionnaire. Overall and subscale scores range from 0 to 100. Lower cores correspond to higher levels of disability (e.g., 0 corresponds to complete disability or responding "extremely" limited, difficult or bothersome to all questions answered), withe a score of 100 corresponds to no disability (e.g., responding "not at all" limited, difficult or bothersome to all questions answered). For Satisfaction questions, a score of 100 corresponds to extreme satisfaction with current treatment.
Quality of Life Health Outcomes using EuroQol-5D-5L | Up to 24 months
  The EQ-5D-5L quality of life questionnaire will be used to assess health related outcomes. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The lower the number, the better the impact on quality of life.
Number of patients with gender association, Atrial fibrillation risk factors and risk factor management | Up to 24 months
  GENESIS PRAXY Gender Questionnaire
Number of patients with recurrent AF Catheter ablations | Up to 60 months
  Any subsequent catheter ablations after the initial procedure
Number of patients with recurrent cardioversions for atrial fibrillation | Up to 60 months
  Electrical or chemical cardioversions
Number of patients with Major bleeding | Up to 60 months
  Fall in Hgb of ≥2 g/dL, transfusion of ≥2 units packed red blood cells (PRBC) or whole blood, in a critical location (e.g., intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial
Number of Deaths | Up to 60 months
  Study Exit due to death from time of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, MD, FRCPC, Principal Investigator — Nova Scotia Health
Locations (7):
- Canada (7):
  - Foothills Hospital, Calgary, Alberta
  - QEIIHSC, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Regina General Hospital, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No